CLINICAL TRIAL: NCT05121038
Title: A Phase 1B/2A Trial of CEND-1 in Combination with Neoadjuvant FOLFIRINOX Based Therapies in Pancreatic, Colon and Appendiceal Cancers (CENDIFOX)
Brief Title: CEND-1 in Combination with Neoadjuvant FOLFIRINOX with or Without Panitumumab
Acronym: CENDIFOX
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anup Kasi (Other)
Collaborators: Cend Therapeutics Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Anup Kasi, MD, MPH, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2021-CENDIFOX
Record Dates: First submitted 2021-10-19; First posted 2021-11-16 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-08

CONDITIONS: Colon Cancer; Pancreas Cancer; Digestive Cancer
MeSH Terms: conditions — Colonic Neoplasms; Pancreatic Neoplasms; Gastrointestinal Neoplasms | interventions — Panitumumab; folfirinox; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 Pancreatic Cancer (Experimental): Biopsy for tissue immune profile if archived tissue not available. Folfirinox infusion for 3 cycles followed by a repeat biopsy for a second tissue immune profiling. Folfirinox plus CEND-1 infusion for 3 cycles. Seventy-two hours after last infusion participant will have surgery.
  Interventions: Drug: CEND-1; Drug: Folfirinox
- Cohort 2 Peritoneal Mets (Experimental): Biopsy for tissue immune profile if archived tissue not available. Folfirinox plus Panitumumab (if RAS/BRAF) infusion for 3 cycles followed by a repeat biopsy for a second tissue immune profiling. Folfirinox plus Panitumumab (if RAS/BRAF positive) and CEND-1 infusion for 3 cycles. Seventy-two hours after last infusion participant will have surgery.
  Interventions: Drug: CEND-1; Drug: Panitumumab; Drug: Folfirinox
- Cohort 3 Oligomets Colon Cancer (Experimental): Biopsy for tissue immune profile if archived tissue not available. Folfirinox plus Panitumumab (if RAS/BRAF) infusion for 3 cycles followed by a repeat biopsy for a second tissue immune profiling. Folfirinox plus Panitumumab (if RAS/BRAF positive) and CEND-1 infusion for 3 cycles. Seventy-two hours after last infusion participant will have surgery.
  Interventions: Drug: CEND-1; Drug: Panitumumab; Drug: Folfirinox

INTERVENTIONS:
Drug: CEND-1 — The treatment with CEND-1 will be given as an intravenous (IV) infusion (through a needle in a vein) at the clinic once every 14 days (or Day 1 of every 14-day cycle starting in Cycle 4).
  Other Names: LSTA1; Certepetide
Drug: Panitumumab — Up to ten (10) participants with cancer that has spread to certain areas of the body and who have a certain gene in the tumor called "RAS/BRAF wild type" will receive another drug called panitumumab in addition to CEND-1 and FOLFIRINOX.
  Arms: Cohort 2 Peritoneal Mets; Cohort 3 Oligomets Colon Cancer
Drug: Folfirinox — FOLFIRINOX is a name for a chemotherapy treatment regimen that includes several different drugs that are given in a certain order.
  All of these drugs are given as an intravenous (IV) infusion (through a needle in a vein) at the clinic once every 14 days (or Day 1 of every 14-day cycle).
  * Oxaliplatin - dose is 85 mg / m2 the infusion takes about 2 hours. then
  * Leucovorin - dose is 400 mg / m2 - this is given at same time with irinotecan (below) and the infusion takes about 1.5 hours.
  * Irinotecan - dose is 180 mg / m2 - this is given at same time with leucovorin (above), and the infusion takes about 1.5 hours.
  then
  • Fluorouracil - dose is 2400 mg / m2 - this infusion takes 46 to 48 hours (2 days) with an IV pump done at home.
  Other Names: Oxaliplatin,Leucovorin,Irinotecan,Fluorouracil

SUMMARY:
This is a phase IB/IIA trial to ensure the safety of Certepetide (LSTA1/CEND-1) in combination with with Folfirinox with or without Panitumumab for treatment of pancreatic, colon and appendiceal cancers

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 - 1
* One or more lesions evaluable on MRI, positive emission tomography (PET)/CT, or dedicated CT scan according to RECIST v1.1
* Patients with histologically confirmed pancreatic ductal adenocarcinomas, colorectal and appendiceal adenocarcinomas
* For cohort 1: Resectable Pancreatic Cancer: No evidence of distant metastasis and tumor mass showing no extension to superior mesenteric artery (SMA) and hepatic artery. There must be clear fat plane between SMA and celiac axis. Patent superior mesenteric vein (SMV/portal vein (PV) with no distortion of venous architecture. Please refer to 2021 NCCN PDAC Guidelines
* For cohort 1: Borderline Resectable Pancreatic Cancer: defined as localized cancer with 1 or more of the following features: "a) an interface between the primary tumor and superior mesenteric vein (SMV)-portal vein (PV) measuring 180o or greater of the circumference of the vein wall, and/or b) short-segment occlusion of the SMV-PV with normal vein above and below the level of obstruction that is amenable to resection and venous reconstruction and/or c) short segment interface of any degree between tumor and hepatic artery with normal artery proximal and distal to the interface that is amenable to resection and arterial reconstruction and/or d) an interface between the tumor and SMA or celiac trunk measuring less than 180o of the circumference of the artery wall. Please refer to 2021 National Comprehensive Cancer Network (NCCN) Pancreatic Ductal Adenocarcinoma (PDAC) Guidelines
* For cohort 2: Peritoneal Metastases due to Colorectal Cancer or Invasive Adenocarcinoma of the Appendix
* For cohort 3: Oligometastatic colorectal cancer: resectable metastases as determined by multidisciplinary evaluation. Patients with bilobar liver metastases or oligometastatic liver and lung metastases that requires resection of one or more metastases are also allowed
* Eligible for treatment with FOLFIRINOX with or without panitumumab
* Life expectancy of at least 3 months
* Adequate archival tissue from prior biopsy for biomarker evaluation or willingness to undergo biopsy before treatment starts and on treatment
* Medically fit to undergo complex major abdominal surgery at end of study treatment
* Women of childbearing potential must have a negative serum pregnancy test within 72 hours prior to enrollment
* Adequate organ function

Exclusion Criteria:

* Simultaneously enrolled in any therapeutic clinical trial
* Concurrent use of any other anti-cancer therapy, including chemotherapy, targeted therapy, immunotherapy, or biological agents
* Prior chemotherapy or any other investigational agents for the treatment of cancer within 2 years prior to enrollment on this study
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Is pregnant or breastfeeding
* Has a known allergic reaction to any excipient contained in the study drug formulation
* Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment
* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
* Known infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the investigator
* Participants with known brain metastases. Screening for brain metastases with head imaging is not required
* History of prior or current synchronous malignancy, except:

  * Malignancy that was treated with curative intent and for which there has been no known active disease for >3 years prior to enrollment
  * Curatively treated non-melanoma skin cancer, cervical cancer in situ, or prostatic intraepithelial neoplasia, without evidence of prostate cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Drug Safety: Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 24 months
  Adverse Events : Counts and proportions of grade 3 -5 Adverse Events

SECONDARY OUTCOMES:
Overall survival (OS) | 48 months
  Overall survival (OS) will be reported using median survival time along with a 90% confidence interval
Disease-free survival (DFS) | 48 months
  Disease-free survival (DFS) will be reported using median survival time along with a 90% confidence interval
Overall response rate (ORR) | 24 months
  Overall response rate (ORR) will be reported as a proportion with 90% confidence interval.
RO resection rate (RORR) | 24 months
  RO resection rate (RORR) will be reported as a proportion with 90% confidence interval.
Pathological response rate (PCR) . | 24 months
  Pathological response rate (PCR) will be reported as a proportion with 90% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Anup Kasi, MD, Principal Investigator — University of Kansas Medical Center
Locations (3):
- United States (3):
  - The University of Kansas Cancer Center (KUCC), Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - The University of Kansas Medical Center, North Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: Undecided